CLINICAL TRIAL: NCT06160817
Title: Effect of Ulcer Location on Debridement Frequency: A Pilot Randomized Controlled Trial Comparing Weekly and Second-weekly Sharp Debridement in Diabetic Foot Ulcers
Brief Title: Ulcer Location and Debridement Frequency: Weekly vs. Biweekly Sharp Debridement in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, FRANCISCO JAVIER ALVARO AFONSO, Associate Professor with a Ph.D, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23/695-EC_X
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot; Wound Heal
Keywords: Diabetes; Diabetic foot ulcer; Sharp wound debridement; wound healing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study employs a prospective, randomized controlled trial design with parallel assignment. The primary objective is to assess the impact of two different debridement modalities, specifically weekly and biweekly sharp debridement, on granulation tissue and healing time in patients with diabetic foot ulcers (DFUs). The study includes three stratified groups based on the location of the ulcer: digital DFUs, DFUs under metatarsal heads, and DFUs in the plantar region of midfoot/heel. Participants meeting inclusion criteria will be randomly assigned to either the weekly or biweekly sharp debridement groups within each location-based stratum. The study aims to elucidate the optimal frequency of debridement based on ulcer location. Outcome measures include the assessment of granulation tissue and healing time. The trial is conducted at the University Podiatry Clinic, and the anticipated duration is from january to april 2024
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind design. The treating clinician, responsible for administering the sharp debridement, is the sole individual aware of the patients' treatment group assignments. Both the participants and the key study personnel, including the principal investigator responsible for data collection and the data analyst responsible for data interpretation, are blinded to the treatment allocation. This approach aims to minimize potential biases and ensure a rigorous evaluation of the effects of weekly and biweekly sharp debridement on granulation tissue and healing time in patients with diabetic foot ulcers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Sharp Debridement (Active Comparator): * Participants in this arm will undergo sharp debridement on a weekly basis.
  * Purpose: Evaluate the effect of weekly sharp debridement, in combination with conventional treatment, on granulation tissue and healing time in diabetic foot ulcers. And assess if this regimen yields better outcomes for ulcers with a specific location.
  * Active Comparator: Yes, as it represents an active treatment modality.
  Interventions: Procedure: Conservative sharp debridement
- Biweekly Sharp Debridement (Active Comparator): * Participants in this arm will undergo sharp debridement on a biweekly basis.
  * Purpose: Assess the impact of biweekly sharp debridement, in combination with conventional treatment, on granulation tissue and healing time in diabetic foot ulcers. And assess if this regimen yields better outcomes for ulcers with a specific location.
  * Active Comparator: Yes, as it represents an active treatment modality.
  Interventions: Procedure: Conservative sharp debridement

INTERVENTIONS:
Procedure: Conservative sharp debridement — The debridement method for all patients, regardless of the assigned sequence, will involve the removal of non-viable tissue from the ulcer bed, edges, and perilesional skin using a scalpel (No. 3) with a No. 10 and/or No. 15 blade, along with Adson forceps and straight dissecting forceps.

SUMMARY:
The goal of this clinical trial is to determine the optimal frequency for sharp debridement in promoting the healing of diabetic foot ulcers (DFUs).

The main questions it aims to answer are:

1. What is the comparative effect of weekly sharp debridement versus biweekly sharp debridement in combination with conventional treatment on granulation tissue and healing time in patients with DFUs?
2. What is the optimal modality or frequency of debridement based on the location of the DFU?

Participants (ulcerated diabetic patients) will:

* Undergo sharp debridement on a weekly basis (Group A).
* Undergo sharp debridement on a biweekly basis (Group B).

Researchers will compare Group A (weekly sharp debridement) with Group B (biweekly sharp debridement ) to see if the frequency of sharp debridement has a significant effect on granulation tissue and healing time in diabetic foot ulcers.

In each group, there will be patients with ulcers in different locations (toes, metatarsal heads, and midfoot/hindfoot) to assess the effect of debridement based on the lesion location

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older who provide written informed consent.
* Patients with Type 1 or Type 2 Diabetes mellitus with a glycated hemoglobin (HbA1c) concentration ≤ 10% (determined in the past 3 months).
* DFUs with the following locations: digital, under metatarsal head, midfoot, and hindfoot.
* DFUs of grades IA, IIA, IB, IIB, IC, IIC, ID, and IID according to the University of Texas Classification.
* DFUs with grades PEDIS 1 - no infection, PEDIS 2 - mild infection, and PEDIS 3 - moderate infection, as per the PEDIS-IDSA classification.
* Neuropathic and neuroischemic ulcers.
* DFUs with grades 0 (absence of ischemia), 1 (mild ischemia), and 2 (moderate ischemia) according to the WIfI (Wound, Ischemia, and foot Infection) Classification, determined by palpation of at least one distal pulse, Ankle-brachial index (ABI) ≥ 0.5, ankle systolic blood pressure ≥ 50 mmHg, or a value ≥ 30 mmHg for toe systolic blood pressure and transcutaneous oxygen pressure (TcpO2).
* Study ulcer surface area between 0.5 cm² and 30 cm² after debridement.
* Duration of the DFU between 2-50 weeks

Exclusion Criteria:

* Patients with severe renal insufficiency requiring dialysis.
* Patients with congestive heart failure (CHF) above Class II, meaning CHF that causes a limitation of physical activity.
* Patients with active coronary disease or a significant adverse cardiac event in the past 18 months, defined as any of the following circumstances: fluctuating symptoms attributed to coronary disease, interventional procedure such as coronary artery bypass grafting or percutaneous coronary intervention (stent placement), worsening of cardiac ejection fraction, increased need for medication used to treat coronary disease, or known presence of coronary lesion with ≥ 70% diameter stenosis that has been previously revascularized.
* Patients with a life expectancy < 6 months.
* Patients with Acquired Immunodeficiency Syndrome (AIDS) or confirmed Human Immunodeficiency Virus (HIV) infection.
* Patients with confirmed diagnosis of hepatitis C virus antibodies or hepatitis C virus surface antigen.
* Pregnant or lactating women, or women of childbearing age not following an effective contraceptive method.
* Patients with critical limb ischemia determined by: Absence of both distal pulses or an ABI ≤ 0.4, ankle systolic blood pressure < 50 mmHg, or a value < 30 mmHg for toe systolic blood pressure and TcpO2, translating to Grade 3 (severe ischemia) according to the WiFi classification.
* DFUs of grades IIIA, IIIB, IIIC, and IIID according to the University of Texas Classification.
* DFUs with PEDIS grades 3O - Moderate infection with osteomyelitis, PEDIS 4 - Severe infection (excluding PEDIS 4O) according to the PEDIS-IDSA classification.
* Patients unable to understand the purposes and objectives of the study.
* Patients with a history of non-compliance with medical treatments (assessed through patient medical history, poor adherence to previous treatments, and therapeutic non-compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Clinical presentation of the ulcer bed | once per week until wound closure, with a maximum follow-up period of 12 weeks
  The clinical presentation of the ulcer bed will be assessed using the Wollina Wound Score, a validated scale designed to comprehensively evaluate various aspects of wound healing.
  The higher the score on this scale, the higher the quality of the wound granulation tissue. The maximum score is 7 points, and the minimum is 0.
  The scale evaluates 3 items to which you assign a score as follows:
  * Presence of granulation tissue in the wound bed: Absence = 0, one-quarter of the ulcer area = 1, half of the area = 2, three-quarters of the area = 3, and complete = 4.
  * Tissue color: Pale = 0, pink = 1, and bright red = 2.
  * Tissue consistency: Spongy = 0, and solid = 1
Healing time | 1 to 12 weeks
  Healing time will be measured (in weeks) as the duration from the initiation of the study intervention until complete closure of the diabetic foot ulcer.

SECONDARY OUTCOMES:
Reduction in ulcer area | Weekly over a period of 12 weeks.
  Change in ulcer area at each follow-up visit compared to the initial measurement. The reduction in ulcer area will be quantified in square centimeters.
Clinical characteristics of the ulcer : Perilesional Skin | Weekly over a period of 12 weeks.
  Assessment of the skin surrounding the ulcer.
  * Intact Skin
  * Erythematous skin
  * Edematous skin
  * Macerated skin
  * Scaly or dry skin
  * Necrotic skin
  * Ecchymotic skin
  * Hyperkeratotic skin
Clinical characteristics of the ulcer: Perilesional Edges | Weekly over a period of 12 weeks.
  Examination of the edges surrounding the ulcer.
  * Healthy edges
  * Dry edges
  * Necrotic edges
  * Hyperkeratotic edges
  * Macerated edges
  * Hyperemic edges
  * Erythematous edges
  * Raised edges
  * Detached edges
Clinical characteristics of the ulcer: Exudate Level | Weekly over a period of 12 weeks.
  * Qualitative measurement: Absent, low, moderate or high
  * Characterization of the wound exudate: serous, sanguineous, purulent, fibrinous and mixed (seropurulent, serosanguineous)
Clinical characteristics of the ulcer: Type of Tissue in the Wound Bed | Weekly over a period of 12 weeks.
  Identification and categorization of the tissue present in the wound bed.
  * Granulation
  * Hypergranulation
  * Slough
  * Necrotic
Clinical characteristics of the ulcer: Local Clinical Signs of Infection | Weekly over a period of 12 weeks.
  Systematic evaluation of any local clinical signs indicating infection.
  * Presence
  * Absence

OTHER OUTCOMES:
SINBAD classification of diabetic foot ulcers | Weekly over a period of 12 weeks.
  Application of the SINBAD (Site, Ischemia, Neuropathy, Bacterial Infection, Area, and Depth) classification system to categorize and characterize diabetic foot ulcers

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Álvaro Afonso, Podiatrist, Principal Investigator — University Podiatry Clinic, "Universidad Complutense de Madrid"
Locations (1):
- Clínica Universitaria Podología, Universidad Complutense, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No